CLINICAL TRIAL: NCT01334710
Title: A Phase II Trial of OSI-906 and Sorafenib in Advanced Hepatocellular Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: safety issue observed on another hepatocellular study using OSI906
Sponsor: Emory University (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Bassel El-Rayes, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047003; WCI1887-10 (Other: Other)
Record Dates: First submitted 2011-04-06; First posted 2011-04-13 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Liver Cancer
Keywords: Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib; 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and OSI-906 (Experimental): This is a single arm phase II trial designed to evaluate the effect of adding OSI-906 to sorafenib in patients with hepatocellular cancer. The study is designed to evaluate the safety of the regimen in the first six patients.
  Interventions: Drug: Sorafenib and OSI-906

INTERVENTIONS:
Drug: Sorafenib and OSI-906 — Sorafenib - 400 mg twice daily OSI-906 - 150 mg twice daily
  Other Names: Nexavar

SUMMARY:
The purpose of this study is to evaluate the effect of combining a new investigational drug (OSI-906) with a standard drug (sorafenib) on the control of liver cancer (hepatocellular cancer). Sorafenib (brand name Nexavar®) is a drug that is approved for the treatment of advanced liver cancer. It works by stopping the growth of new blood vessels around the tumor. OSI-906 is an investigational agent that works by inhibiting the effects of a growth hormone on the cancer. The safety and efficacy of combining OSI-906 and sorafenib in the treatment of liver cancer risk not known. The current study will confirm the safety of the combination in the first six patients and evaluate the activity of the combination in patients with advanced liver cancer.

In addition, the study will aim at collecting blood samples from patients to evaluate the level of OSI-906 in patients receiving the combination of the two drugs. The study also will collect samples of the tumor to evaluate for markers that can predict in which patient the combination is effective.

DETAILED DESCRIPTION:
The purpose of the trial is first to evaluate the safety of the combination of OSI-906 and sorafenib in patients with hepatocellular cancer (HCC). Patients will be treated in groups of three with full dose sorafenib and OSI-906. If we do not observe any significant side effects, then three additional patients will be treated at the same dose level. After confirming the safety of the combination (possibly after first six patients) the study will proceed with regular accrual. The patients will receive the treatments orally and will be evaluated by physical exam, blood work and imaging. If the cancer is well controlled and the therapy is well tolerated then patients will continue on the trial. If the side effects are significant or the tumor starts to grow or the patients wishes to stop therapy the patient at that time will be taken off trial.

The trial will collect blood samples to evaluate the level of the investigational agent in the blood. Also samples of the patients tumor will be analyzed to evaluate for markers that may predict who benefits from treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable, histological diagnosis of HCC and whose disease is not amenable to surgical or regional therapy.
* Prior allowed therapy: surgery, regional therapy (if more than 6 weeks have elapsed from therapy and if there is an indicator lesion outside the treated area or if there is clear evidence of progression in the treated lesion), or adjuvant sorafenib (if disease relapsed more than 6 months after completion of adjuvant therapy).
* Patient with cirrhosis must have Childs-Pugh score of either A or B7.
* Performance status of 0-2.
* Organ function requirements: hemoglobin > 9.0mg/dl; granulocyte count > 1,000 /mm³ , platelets > 40,000/mm³ , alanine aminotransferase (ALT)/aspartate aminotransferase (AST) up to 5 times the institutional upper limit of normal, alkaline phosphatase < 4 times the institutional upper limit of normal and serum creatinine < 2mg/dl.
* Patients must provide verbal and written informed consent to participate in the study.
* Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Exclusion Criteria:

* Patients with mixed histology or fibrolamellar variant.
* Fasting glucose >150 mg/dl and any prior history of diabetes.
* Patients with Type 1 diabetes mellitus or Type 2 diabetes mellitus currently requiring insulinotropic or insulin therapy.
* Prior systemic therapy for metastatic disease.
* Corrected QT (QTc) interval > 450 msec at baseline.
* Concomitant drugs that prolong the QTc interval.
* Significant cardiac disease defined as: congestive heart failure (NYHA class 2 or higher) or active coronary artery disease (MI within 6 months of study enrollment).
* Pregnant or breast-feeding females.
* Serious active infections.
* Encephalopathy.
* Uncontrolled ascites defined as symptomatic ascites not controlled with diuretic treatments.
* Active second primary malignancy except for is situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin within less than one year of enrollment into the study.
* Use of drugs that have a known risk of causing Torsades de Pointes (TdP) are prohibited within 14 days prior to enrollment.
* Use of the potent CYP1A2 inhibitors such as ciprofloxacin and fluvoxamine. Other less potent CYP1A2 inhibitors/inducers are not excluded.
* Patients with a history of poorly controlled gastrointestinal disorders that could affect the absorption of study drug (e.g., Crohn's disease, ulcerative colitis, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bassel El-Rayes, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib and OSI-906: This is a single arm phase II trial designed to evaluate the effect of adding OSI-906 to sorafenib in patients with hepatocellular cancer. The study is designed to evaluate the safety of the regimen in the first six patients.
  Sorafenib and OSI-906 : Sorafenib - 400 mg twice daily OSI-906 - 150 mg twice daily
Period: Overall Study
Arm/Group | Sorafenib and OSI-906
Started | 3
Completed | 0 (Due to safety signals in a parallel trial ON OSI906 in hepatocellular cancer the trial was stopped.)
Not Completed | 3
Not completed — Trial was terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib and OSI-906
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Comparison of MRI/CT Scans to Pre-treatment Scan
Description: Efficacy will be measured by evaluating the number of patients who do not have disease progression (measured by CT or MRI scan) 5 months after starting treatment. Assessment of the endpoint of disease progression will be performed every 2 months using either CT or MRI scan. Participants will remain on the study until either evidence of disease progression or unacceptable side effects develop. This period is expected to be on the average 6 months long.
Time Frame: 6 months
Population: Trial was terminated early.
Arm/Group | Sorafenib and OSI-906
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity Assessment
Description: Evaluate the proportion of participants treated with OSI-906 and sorafenib who develop serious adverse events.
Time Frame: 28 days from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib and OSI-906
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib and OSI-906
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
A second trial evaluating OSI906 in hepatocellular cancer was being run in parallel to this trial. There were safety signals in the second trial which led to stopping this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes